CLINICAL TRIAL: NCT03009604
Title: Does Simethicone Improve Operative Field in Gynecological Operations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Altayeb Abd alal Mostafa Mohammad, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIM
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Benign Gynecologic Neoplasm
MeSH Terms: interventions — Simethicone; Enema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simethicone (Experimental): women take 6 tablets (2 tablets after each meal) and to fast overnight before the operation
  Interventions: Drug: Simethicone
- Enema (Active Comparator): women take 3 rectal Enema (8:00 pm, 12:00 am & 8:00 am) and to fast over night before the operation.
  Interventions: Drug: Enema

INTERVENTIONS:
Drug: Simethicone — Simethicone 40mg oral tablets
  Arms: Simethicone
Drug: Enema — sodium dihydrogen phosphate dihydrate 19.2 gram & disodium hydrogen phosphate dodecahydrate 7.2 gram, in addition to purified water
  Arms: Enema

SUMMARY:
Mechanical bowel preparation aims to decrease the volume fecal content in the colon, which thereby decreases the total colony count of bacteria, thus, decreasing peritoneal contamination in case of bowel injury, improving the access to the surgical field and facilitating intraoperative bowel manipulation

ELIGIBILITY:
Inclusion Criteria:

Gynecological operations for benign conditions as hysterectomy, ovarian cystectomy and myomectomy.

Exclusion Criteria:

1. History of allergic reaction to study drugs.
2. More than one scar of previous operation.
3. Suspicious of malignancy.
4. Psychiatric disorders.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
the degree of small & large bowel preparation | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided